CLINICAL TRIAL: NCT00696033
Title: Exploring the Effects of Diazepam and Lorazepam on the Neural Correlates of Perceptual Priming and Explicit Memory in Healthy Volunteers
Brief Title: Exploring the Effects of Diazepam and Lorazepam
Acronym: ibid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 3777
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2009-09

CONDITIONS: Healthy Subjects
Keywords: Benzodiazepines; Lorazepam; Diazepam; Memory; Perceptual priming; Functional brain imaging; FMRI
MeSH Terms: interventions — Diazepam; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Oral Lorazepam
  Interventions: Drug: Lorazepam
- 2 (Experimental): Oral Diazepam
  Interventions: Drug: Diazepam
- 3 (Placebo Comparator): Oral placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Diazepam — Diazépam drug (0,3 mg/kg) on a single oral intake
  Arms: 2
Drug: Lorazepam — Lorazépam drug (0,038 mg/kg) on a single oral intake
  Arms: 1
Drug: placebo — lorazépam placebo or Diazépam placebo
  Arms: 3

SUMMARY:
Aims :

* exploring lorazepam (0.038 mg/kg) effects, after a single oral intake, in healthy volunteers, on the neural correlates of encoding and retrieval of information during a word-stem completion task (implicit memory), using fMRI
* comparing lorazepam effects to diazepam (0.3 mg/kg)effects
* exploring benzodiazepines effects, after a single oral intake, on the neural correlates of successful encoding of information within explicit memory using fMRI

Hypothesis :

* both diazepam and lorazepam will impair explicit memory performance, but lorazepam only will impair perceptual priming
* lorazepam and diazepam will modify the normal correlates of information encoding within explicit memory
* lorazepam only will alter the neural correlates of perceptual priming

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between 18 and 30 years
* Students in medicine, dentistry or pharmacy
* French as a mother language

Exclusion criteria:

* Medical condition influencing brain function (neurological or psychiatric)
* Asthma
* General anesthesia in the 3 last months
* Drug addiction (DSM IV criteria)
* Regular medical treatment (except contraceptive pill)
* Significant impairment observed during a medical examination including ECG
* Intake of any psychotropic drug that can have a effect during testing
* IQ (Wechsler) < 100
* FMRI contra-indication (implantable magnetic material, claustrophobia)
* Known allergy to benzodiazepine or lactose
* > 10 cigarettes/day
* Pregnant or breast-feeding woman
* No health insurance
* Subjects who do not complete the entire study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Exploring lorazepam (0.038 mg/kg) effects, after a single oral intake, in healthy volunteers, on the neural correlates of encoding and retrieval of information during a word-stem completion task (implicit memory), using fMRI | After a single oral intake

SECONDARY OUTCOMES:
Comparing lorazepam effects to diazepam (0.3 mg/kg)effects | After a single oral intake
Exploring benzodiazepines effects, after a single oral intake, on the neural correlates of successful encoding of information within explicit memory using fMRI | After single oral intake

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Vidailhet, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Centre d'investigation clinique, hôpital civil, Strasbourg
  - Clinique psychiatrique, hôpital civil, Strasbourg